CLINICAL TRIAL: NCT01802944
Title: Intranasal Insulin: A Novel Treatment for Gulf War Multisymptom Illness
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bronx Veterans Medical Research Foundation, Inc (Other)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency); Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GW110054
Record Dates: First submitted 2013-02-19; First posted 2013-03-04 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Chronic Multisymptom Illness in Gulf War Veterans

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10 IU BID (Experimental): 10 IU BID Intranasal Insulin
  Interventions: Drug: Intranasal Insulin
- 20 IU BID (Experimental): 20 IU BID Intranasal Insulin
  Interventions: Drug: Intranasal Insulin
- PLACEBOS (Experimental): Saline nasal solution used as placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Intranasal Insulin
  Arms: 10 IU BID; 20 IU BID
Drug: Placebos
  Arms: PLACEBOS

SUMMARY:
Following their deployment to the 1991 Gulf War, many veterans (GWV) reported a constellation of unexplained health symptoms; common among them were attention and memory difficulties, fatigue, joint pain, headaches, gastrointestinal complaints, and mood and sleep problems. Despite the passage of time, the symptom complex persists for many veterans. Indeed, it is estimated that at least 25 percent of GWV (nearly 170,000 veterans) have a persistent form of chronic multisymptom illness (CMI). GW deployed veterans are also developing significantly more chronic diseases such as diabetes, hypertension, arthritis, and coronary heart disease than their non-deployed veteran peers putting these individuals at risk for accelerated aging-related diseases of the peripheral and central nervous system (CNS). Recent studies have shown a slowing of response speed that affects mental flexibility across multiple cognitive domains (memory, attention, visuospatial functions) especially on tests that were timed and computerized and where small differences in cognitive reaction times could be measured. Recent studies also have suggested that the response inhibition deficits shown in GWV may reflect executive system dysfunction as reflected by slower motor responses across multiple cognitive domains.

To date, there are no treatments that have been shown to improve the health or cognitive difficulties of GW veterans; thus there is an urgent need to establish effective, safe, and tolerable treatments for GW CMI. Previous studies in other cognitive disorders have found that intranasal insulin improves memory, attention, and mood, reduces neuroinflammation, and modulates cortisol levels; it has also been identified as a treatment that has the capacity to alter many of the leading problems of GW CMI.

During this study there are 2 treatment groups and a placebo group that will last for 8 weeks. The treatment groups will self-administer their designated dosage of insulin through a nasal pump twice a day, while the placebo group will administer saline through a nasal pump twice a day. These doses have been shown to be effective and safe. The primary outcome measure will assess improvements in verbal delayed memory using a specific list learning task and on a measure of selective attention. The study will assess improvements in overall physical health and mood by asking the participants to complete self report questionnaires. Neuroendocrine measures will also be obtained in order to evaluate changes in glucose, insulin, and cortisol levels and examine their impact on GW CMI.

Intranasal insulin has shown great promise in improving memory, attention, and mood in both older adults with cognitive impairment as well as normal subjects. Thus, this proposal could prove intranasal insulin to be an effective, safe, and affordable therapy for these ailing veterans.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a veteran of the 1991 Gulf War.
* Veteran meets criteria for chronic multisymptom illness based Kansas Gulf War Study (Steele, 2000) criteria and must meet criteria in the cognitive symptom domain.

Exclusion Criteria:

* Veteran lacks the capacity to provide consent.
* Veteran has diabetes, a major medical or neurological disorder or moderate-severe traumatic brain injury.
* Veteran has a history of hypoglycemia.
* Veteran is taking oral or nasal corticosteroids, insulin or oral hypoglycemic agents.
* Veteran has an irregular nasal cavity (i.e. nasal polyps etc.) or is using nasal sprays on a regular basis.
* Veteran has a lifetime diagnosis of schizophrenia, schizoaffective disorder or type I bipolar disorder.
* Veteran is at high risk from a mental perspective as evidence by having been psychiatrically hospitalized or attempted suicide within the previous 2 years or has current active suicidal ideation.
* Veteran is pregnant or breastfeeding or plans to become pregnant within the year.

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Memory Functioning | Eight weeks
  To assess the efficacy of two different doses (10 IU BID and 20 IU BID) of daily intranasal insulin for eight weeks on memory functioning in Gulf War Veterans with Chronic Multisymptom Illness. The primary clinical outcome measure will be a change in the performance on the delayed verbal memory score on a list learning task (California Verbal Learning Test (CVLT). To determine the sustainability of change in cognitive status, the response from treatment endpoint (end of 8-week treatment period) to one month follow-up (post end of 8-week treatment period) will also be assessed for the primary outcome measure.
Attention Functioning | Eight Weeks
  To assess the efficacy of two different doses (10 IU BID and 20 IU BID) of daily intranasal insulin for eight weeks on attention functioning in Gulf War Veterans with Chronic Multisymptom Illness. The primary clinical outcome measure will be a change in performance on a selective attention task (Stroop Color-Word Interference Task) from treatment baseline to endpoint. To determine the sustainability of change in cognitive status, the response from treatment endpoint (end of 8-week treatment period) to one month follow-up (post end of 8-week treatment period) will also be assessed for the outcome measure.

SECONDARY OUTCOMES:
Physical Health | Eight weeks
  An outcome measure will be the changes in physical health over the course of active treatment. The primary measure of physical health will be the Physical Components Score (PCS) from the Standard Form 12-veteran version (SF-12V). The clinical outcome measure will be the change in PCS score from treatment baseline to endpoint. To determine the sustainability of change in PCS scores, the response from treatment endpoint to one month follow-up will also be assessed.
Mood | Eight Weeks
  An outcome measure will be the changes in mood over the course of active treatment. The primary measure of mood will be obtained from the Profile of Mood States (POMS) vigor scale. The clinical outcome measure will be the change in POMS scores from treatment baseline to endpoint. To determine the sustainability of change in POMS scores, the response from treatment endpoint to one month follow-up will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Golier, MD, Principal Investigator — Chief of Psychiatry Bronx VA Medical Center
Locations (2):
- United States (2):
  - VA Boston Healthcare System, Boston, Massachusetts
  - James J. Peters VA Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Undecided